CLINICAL TRIAL: NCT03576352
Title: Pediatric Emergency Front of the Neck Access (eFONA): Assessing a Novel Experiential Learning Approach
Brief Title: Emergency Front of the NecK Access (eFONA) in Children
Acronym: eFONA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: Riva-Ulmer2017
Record Dates: First submitted 2018-06-18; First posted 2018-07-03 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Pediatric Anesthesia; Intubation;Difficult

STUDY DESIGN:
Intervention Model Description: Anesthesiologist, pediatric intensivists, surgeons, and emergency physicians who are most likely to need to perform FONA in small children, shall learn to perform RST emergent pediatric tracheotomy in less than 60 seconds. The investigators seek to measure and study their learning curves for establishing an artificial airway using the RST.
  Single-center interventional trial. The only inclusion criterion is informed consent. A high quality instructional video demonstrating the RST on a rabbit cadaver will teach the participants. Performance time will be defined (from touching the skin until ventilation of the trachea with a standard self-inflating bag connected to the tube).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pediatric anesthesiologist (Experimental): 10 rapid sequence tracheostomy (RST) on rabbit cadaver
  Interventions: Other: a rapid sequence tracheostomy (RST) on rabbit cadaver
- Pediatric intensivists (Experimental): 10 rapid sequence tracheostomy (RST) on rabbit cadaver
  Interventions: Other: a rapid sequence tracheostomy (RST) on rabbit cadaver
- Pediatric surgeons (Experimental): 10 rapid sequence tracheostomy (RST) on rabbit cadaver
  Interventions: Other: a rapid sequence tracheostomy (RST) on rabbit cadaver
- Pediatric emergency physicians (Experimental): 10 rapid sequence tracheostomy (RST) on rabbit cadaver
  Interventions: Other: a rapid sequence tracheostomy (RST) on rabbit cadaver

INTERVENTIONS:
Other: a rapid sequence tracheostomy (RST) on rabbit cadaver — The Rapid Sequence Tracheostomy (RST) consists of the following steps:
  1. Orientational palpation and vertical midline skin incision followed by separation of the strap muscles
  2. Exposure of the trachea and cricoid followed by anterior luxation of the trachea with a Backhaus towel clamp
  3. Perform a vertical puncture with a tip scissors between the Cricoid and 1st tracheal ring followed by a vertical incision of no more than 2 rings in length.
  4. An age adapted tracheal tube is inserted into the trachea and the lungs are ventilated.

SUMMARY:
Study participants will be shown an illustrated training video demonstrating and explaining the RST. The video may be reviewed until the participant feels confident to perform procedure.

The Rapid Sequence Tracheostomy (RST) consists of the following steps:

1. Orientational palpation and vertical midline skin incision followed by separation of the strap muscles
2. Exposure of the trachea and cricoid followed by anterior luxation of the trachea with a Backhaus towel clamp
3. Perform a vertical puncture with a tip scissors between the Cricoid and 1st tracheal ring followed by a vertical incision of no more than 2 rings in length.
4. An age adapted tracheal tube is inserted into the trachea and the lungs are ventilated.

Teaching methodology: Prior to the hands-on training of eFONA, all participants shall watch a 2-minute training video of RST performed on rabbit cadaver following the steps outlined above. During video demonstration, no additional explanation or support will be provided.

Once study participants express confidence to perform the skill, participants shall attempt to perform the RST 10 times. During the RST procedure no additional explanation or support will be provided. Study participants will be allowed to watch the video again between attempts, if needed. Each attempt will be video recorded and time recorded for rater analysis, as outlined above. Successful tracheotomy is defined as ventilation of the lungs by way of a standard self-inflating bag that is to be connected to the tracheal tube or visual confirmation of the tube being placed at least 2 cm inside the trachea (dissection of the rabbit cadaver performed by assistant).

DETAILED DESCRIPTION:
Current difficult airway algorithms end with the need for tracheal airway access to be obtained via Front Of Neck Access (FONA) to achieve oxygenation. In children < 8 years existing recommendations and the literature do not offer guidance on how to perform emergent FONA. Emergent tracheotomy is the potentially life-saving procedure - which needs to be performed without delay. When emergent tracheotomy is attempted in children < 8 years of age, there is a substantial risk for complications. As a result, health care providers who do not have routine at performing this procedure are often reluctant to perform FONA, Diameters, vertical/horizontal dimensions, vocal cord distance, larynx position, and cricothyroid membrane size of the rabbit airway suggest considerable similarities with infant airways, making it a good model to learn this technique. The FONA rapid sequence technique (RST) is a simple technique suitable for emergent pediatric tracheotomy. RST outlines 4 clearly defined steps, that enable airway establishment.

Step 1: Vertical midline skin incision and separate the strap muscles Step 2: Expose trachea and cricoid through palpation, lift and immobilize trachea with a clamp Step 3: Vertical trachea incision with the sharp tip scissors (2 cm) Step 4: Open the trachea and insert the tube The steps are easy to perform, if sufficiently practiced. Anesthesiologist, pediatric intensivists, surgeons, and emergency physicians who are most likely to need to perform FONA in small children, shall learn to perform RST emergent pediatric tracheotomy in less than 60 seconds. The investigators seek to measure and study learning curves of participants for establishing an artificial airway using the RST.

Hypothesis: After having practiced the procedure 10 times, 80% of study participants will not be able to successfully demonstrate FONA within 60 seconds. Alternative hypothesis: study participants will be able to successfully demonstrate FONA within 60 seconds.

Single-center interventional trial. The only inclusion criterion is informed consent. A high quality instructional video demonstrating the RST on a rabbit cadaver will teach the participants. Performance time will be defined (from touching the skin until ventilation of the trachea with a standard self-inflating bag connected to the tube). The investigators seek to assess the learning curves of participants.

Sample size. In order to obtain a lower limit of the 95% Confidence interval of 80% success in FONA the investigators would need 40 study participants assuming 2 failures by the 10th attempt. Statistical methods: Descriptive statistics for demographics. To establish the learning curve the increase over the 3 attempts will be analyzed by repeated ANOVA or Friedman.

For the reasons outlined above the investigators will provide a suitable and valid training model for pediatric airway practitioners to practice the invasive front of neck access technique.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria are informed consent, no previous experience in FONA.

Exclusion Criteria:

none

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-11-10 (Actual); Study Completion 2018-12-23 (Actual)

PRIMARY OUTCOMES:
Performance time | 60 seconds
  The primary outcome will be performance time of RST representing the time from touching the skin until ventilation of the trachea (visualized by lung expansion) indicating the artificial airway as established. Performance time will yield learning curves. The declared intention is to perform RST in less than 60 seconds. Failed/aborted RST will be registered as a 5-minute attempt

SECONDARY OUTCOMES:
Number of attempts | 1 hour
  Number of attempts to perform the skill in <60 s
Number of attempts for plateau | 1 hour
  Number of attempts to reach a time plateau
Preparation of the trachea | 60 seconds
  Time to vertical incision of the trachea with the sharp tip scissors
Vertical incision | 60 seconds
  Time to vertical incision of the trachea with the sharp tip scissors
Training | 1 hour
  Number of times that training video was watched
Suitability | 1 hour
  The subjective rating of the suitability of the given training model

CONTACTS AND LOCATIONS:
Overall Officials: Greif Robert, Prof., Study Chair — Department Anesthesia and Pain Therapy, University Hospital Bern
Locations (1):
- University Hospital Bern, Bern, Switzerland

REFERENCES:
- [Derived] Ulmer F, Lennertz J, Greif R, Butikofer L, Theiler L, Riva T. Emergency front of neck access in children: a new learning approach in a rabbit model. Br J Anaesth. 2020 Jul;125(1):e61-e68. doi: 10.1016/j.bja.2019.11.002. Epub 2019 Dec 4. PMID 31812268